CLINICAL TRIAL: NCT03729375
Title: The Effect Of An Anesthetic Procedure On Post Operative Pain Management In Carpal Tunnel Release
Acronym: CTR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Francisco Schwartz-Fernandes, Assistant Professor, USF College of Medicine, Orthopaedics, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00033480
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Pain, Postoperative; Carpal Tunnel Syndrome
MeSH Terms: conditions — Pain, Postoperative; Carpal Tunnel Syndrome | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10cc Patients (Experimental): Intervention: Group 1 will receive 10cc of intra-operative intra-carpal tunnel anesthetic injection (bupivacaine/Marcaine). Postoperatively, patients will also be prescribed an opioid pain medication in congruence with current standard medical practice. Patients will be contacted at 24-hours, 48-hours, 72-hours, and at 2-week clinic follow-up by research staff and evaluated for pain levels through the LIKERT scale.
  Interventions: Drug: 10cc injection of bupivacaine
- 20cc Patients (Active Comparator): Intervention: Group 2 will receive 20cc of intra-operative intra-carpal tunnel anesthetic injection (bupivacaine/Marcaine). Postoperatively, patients will also be prescribed an opioid pain medication in congruence with current standard medical practice. Patients will be contacted at 24-hours, 48-hours, 72-hours, and at 2-week clinic follow-up by research staff and evaluated for pain levels through the LIKERT scale.
  Interventions: Drug: 20cc injection of bupivacaine

INTERVENTIONS:
Drug: 10cc injection of bupivacaine — 10cc intra-operative injection of bupivacaine into the carpal tunnel of the operative hand/wrist
  Other Names: Bupivacaine (Marcaine)
  Arms: 10cc Patients
Drug: 20cc injection of bupivacaine — 20cc intra-operative injection of bupivacaine into the carpal tunnel of the operative hand/wrist
  Other Names: Bupivacaine (Marcaine)
  Arms: 20cc Patients

SUMMARY:
Carpal Tunnel Syndrome patients undergoing carpal tunnel release surgery performed by the PI will receive intra-operative injections of bupivacaine (Marcaine). Two groups of patients will be randomly selected and will receive either 10cc or 20cc of injection. Their post-operative pain scores and usage of post-operative pain medication will be recorded and analyzed.

DETAILED DESCRIPTION:
This randomized control trial will be conducted at the USF Department of Orthopaedics at the USF Health Morsani Center after receiving approval from the USF Institutional Review Board. Patients will be evaluated Carpal Tunnel Syndrome and screened as candidates for Carpal Tunnel Release surgery, following the inclusion and exclusion criteria. The Medical Record Number (MRN) will be used to randomly assign into treatment interventions. Group 1 and group 2 will receive 10cc and 20cc of intra-operative intra-carpal tunnel anesthetic injection, respectively. Postoperatively, patients will be prescribed an opioid pain medication in congruence with current standard medical practice. Patients will be contacted at 24-hours, 48-hours, 72-hours, and at 2-week clinic follow-up by research staff and will be evaluated for pain levels through the LIKERT scale and pain management through use of prescribed and supplemental pain medications. All data will be analyzed through SPSS v25.

ELIGIBILITY:
Inclusion Criteria:

* patient must be undergoing carpal tunnel release surgery performed by PI
* EMG or Ultrasound diagnosed carpal tunnel syndrome

Exclusion Criteria:

* co-musculoskeletal injuries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-10-04 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
Change in Pain Level in various stages of the post-operative period | Changes in pain scores at 24 hours, 48 hours, 72 hours, and 2 weeks post-operatively
  The investigator will implement a survey using a LIKERT scale regarding post-operative pain levels.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Schwartz-Fernandes, MD, Principal Investigator — USF Orthopaedics
Locations (1):
- University of South Florida Department of Orthopaedics, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No